CLINICAL TRIAL: NCT03270475
Title: Effect of Exercise Training on Skeletal Muscle Proteome Signature of Young Men
Brief Title: Effect of Exercise on Muscle Proteome Signature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morten Hostrup, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Hostrup, PhD, Assistant Professor, PhD, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ACE
Record Dates: First submitted 2017-08-28; First posted 2017-09-01 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): 12-15 training sessions of 30 min over 4-5 weeks
  Interventions: Other: exercise training

INTERVENTIONS:
Other: exercise training — subjects complete 4-5 weeks of training

SUMMARY:
The aim of the study is to investigate skeletal muscle proteome signature changes induced by exercise training in young men

DETAILED DESCRIPTION:
Advances in omics technologies have allowed for the identification of biomarkers with importance for the beneficial adaptations imposed by exercise training. Skeletal muscle exhibits remarkable plasticity to exercise training, as illustrated by pronounced alterations to the proteomic landscape, such as mitochondrial biogenesis. However, despite recent advances that have helped describe the proteomic landscape in response to a period of exercise training, our understanding of the processes pertaining to post-translation modification is scant. In this study, we aim to investigate the human acetylome and proteome in response to exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* VO2max of 45-55 ml/kg/min (+/- SD) / 3000-4000 ml/min (+/- SD)
* Body mass index (BMI) of 19-26 kg/m2
* Normal ECG (electrocardiography)

Exclusion Criteria:

* Serious adverse effects to exercise
* Chronic disease

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle proteome signature | Change from baseline proteome signature at 5 weeks
  proteomics

OTHER OUTCOMES:
Skeletal muscle acetylome signature | Change from baseline acetylome signature at 5 weeks
  acetylomics
Skeletal muscle mitochondrial respiration | Change from baseline at 5 weeks
  Mitochondrial respiratory capacity
Maximal oxygen uptake | Change from baseline at 5 weeks
  Maximal oxygen uptake

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided